CLINICAL TRIAL: NCT06394765
Title: 5-minute Mindful Pain Management Strategy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Adam Hanley, Associate Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00005027
Record Dates: First submitted 2024-04-29; First posted 2024-05-01 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Pain; Chronic Pain; Musculoskeletal Pain
MeSH Terms: conditions — Pain; Chronic Pain; Musculoskeletal Pain

STUDY DESIGN:
Intervention Model Description: This project is a single-site, two-arm, pilot study assessing the feasibility and preliminary efficacy of a 5-minute Mindful Mapping intervention for adults with chronic musculoskeletal pain relative to a time- and attention-matched control condition.
Who Masked: Participant
Masking Description: Participants will be randomized (1:1) using a computer-generated randomization sequence created by the PI prior to the study start date.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindful Mapping (Experimental)
  Interventions: Behavioral: Mindful Mapping
- Serial Sevens (Active Comparator)
  Interventions: Behavioral: Serial Sevens

INTERVENTIONS:
Behavioral: Mindful Mapping — Participants in the Mindful Mapping condition will receive a 5-minute, therapist-guided mindfulness intervention for chronic pain. During this training they will learn the 30-second Mindful Mapping technique, which they will be instructed to use each time they experience a painful sensation over the next 2 weeks. The Mindful Mapping technique consists of focusing on five basic characteristics (shape, weight, density, temperature, movement) of the most intense sensation in the body as it emerges in the present moment while remaining equanimous, i.e., preventing the learned reaction.
  Arms: Mindful Mapping
Behavioral: Serial Sevens — Participants in the control condition will receive a 5-minute, therapist-guided "serial sevens" intervention for chronic pain. During this training, participants will be instructed that each time they experience pain, they will count backwards in their heads by 7 from 100 for 30 second.
  Arms: Serial Sevens

SUMMARY:
This project is a single-site, two-arm, pilot study assessing the feasibility and preliminary efficacy of a 5-minute Mindful Mapping intervention for adults with chronic musculoskeletal pain (n=60) relative to a time- and attention-matched control condition.

DETAILED DESCRIPTION:
This was a two-arm (Mindful Mapping vs. Serial Sevens), remotely delivered, parallel-group, pilot RCT. All procedures were approval by the local IRB and preregistered (NCT06394765). Written informed consent was obtained from all participants prior to their inclusion in the study. Participants were randomly assigned (1:1) to either the Mindful Mapping intervention (n=30) or a control condition, Serial Sevens (n=30). Randomization was performed using a computer-generated sequence.

ELIGIBILITY:
Inclusion Criteria:

* having a chronic pain diagnosis
* being able not to commit to another (new) treatment during the course of the study
* understanding English instructions fluently
* Being 18 and above

Exclusion Criteria:

* having learned to practice mindfulness meditation any time in the past
* being unable to perform most basic tasks due to pain or pain treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-06-13 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Recruitment Feasibility | 3 months
  Examine recruitment rates during the 3 months planned for recruitment.
Randomization Feasibility | 3 months
  Examine randomization rates during the 3 months planned for recruitment.
Intervention Adherence | 5 minutes
  Examine the percentage of participants completing their 5-minute intervention session
Therapeutic Skill Use Adherence | 2 weeks
  Examine the frequency of therapeutic skill use during the 2-week, post-intervention, self-management period.

SECONDARY OUTCOMES:
Treatment Acceptability | Completed at 2- and 6-week follow-ups
  Treatment acceptability will be assessed with the Treatment Acceptability and Preference (TAP) scale. Scores range from 0 to 4, with higher scores reflecting greater acceptability.
Global Impression of Change | Completed at 2- and 6-week follow-ups
  Treatment related improvement will be assessed with the Patient Global Impression of Change scale. Scores range from 0 to 7, with higher scores reflecting greater treatment related improvement.

OTHER OUTCOMES:
Acute Pain Unpleasantness | Will be completed immediately before and after the 5-minute intervention session
  Change in acute pain unpleasantness will be measured with an individual item ("How unpleasant is your pain, right now?") rated on a numeric rating scale. Scores range from 0 to 10, with higher scores reflecting greater acute pain unpleasantness.
Acute Pain Intensity | Will be completed immediately before and after the 5-minute intervention session
  Change in acute pain intensity will be measured with an individual item ("How much pain do you have, right now?") rated on a numeric rating scale. Scores range from 0 to 10, with higher scores reflecting greater acute pain intensity.
Daily Pain Intensity | Daily for 6 weeks
  Change in daily pain intensity from from the first post-intervention day through the 6-week follow-up will be assessed with the pain intensity item from the Pain, Enjoyment, and General Activity scale. Scores range from 0 to 10, with higher scores reflecting greater pain intensity.
Daily Pain Interference | Daily for 6 weeks
  Change in daily pain interference from from the first post-intervention day through the 6-week follow-up will be assessed with the two pain interference items from the Pain, Enjoyment, and General Activity scale. Scores range from 0 to 10, with higher scores reflecting greater pain interference.
Chronic Pain | Baseline, 2 weeks post-treatment, 6 week post-treatment
  Change in chronic pain from baseline through 6-week follow-up will be assessed with the Pain, Enjoyment, and General Activity scale. Scores range from 0 to 10, with higher scores reflecting greater chronic pain.
Physical Function | Baseline, 2 weeks post-treatment, 6 week post-treatment
  Change in physical function from baseline through 6-week follow-up will be assessed with the PROMIS Physical Functioning Short Form. Scores range from 6 to 30, with higher scores reflecting greater physical function.
Sleep | Baseline, 2 weeks post-treatment, 6 week post-treatment
  Change in sleep from baseline through 6-week follow-up will be assessed with the PROMIS Sleep Disturbance Short Form. Scores range from 6 to 30, with higher scores reflecting worse sleep.
Pain Catastrophizing | Baseline, 2 weeks post-treatment, 6 week post-treatment
  Change in pain catastrophizing from baseline through 6-week follow-up will be assessed with the Pain Catastrophizing Scale. Scores range from 0 to 52, with higher scores reflecting greater pain catastrophizing.
Depression | Baseline, 2 weeks post-treatment, 6 week post-treatment
  Change in depression from baseline through 6-week follow-up will be assessed with the Patient Health Questionnaire-2. Scores range from 0 to 6, with higher scores reflecting greater depression.
Anxiety | Baseline, 2 weeks post-treatment, 6 week post-treatment
  Change in anxiety from baseline through 6-week follow-up will be assessed with the Generalized Anxiety Disorder 2-item. Scores range from 0 to 6, with higher scores reflecting greater anxiety.
Prescription Pain Medication Use | Baseline, 2 weeks post-treatment, 6 week post-treatment
  Change in prescription pain medication misuse from baseline through 6-week follow-up will be assessed with the PROMIS Prescription Pain Medication Misuse Short Form. Scores range from 7 to 35, with higher scores reflecting greater medication misuse.
Mindful Pain Management | Baseline, 2 weeks post-treatment, 6 week post-treatment
  Change in the use of mindfulness for pain management from baseline through 6-week follow-up will be assessed with the Mindful Reappraisal of Pain Scale. Scores range from 0 to 54, with higher scores reflecting greater mindful pain management.

CONTACTS AND LOCATIONS:
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No